CLINICAL TRIAL: NCT03852693
Title: Distant Metastases and Long-Term Survival After Complete Resection of Neuroendocrine Tumors of the Appendix: An International Multicenter Study
Brief Title: Distant Metastases and Long-Term Survival After Complete Resection of Neuroendocrine Tumors of the Appendix
Acronym: SurvivApp
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: SurvivApp
Record Dates: First submitted 2019-02-20; First posted 2019-02-25 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Neuroendocrine Tumors of the Appendix

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Tissue blocks of deceased or distant metastatic patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Group
  Interventions: Other: Histopathological review
- Prospective Group
  Interventions: Other: Histopathological review

INTERVENTIONS:
Other: Histopathological review — Histopathological review

SUMMARY:
The aim of the present project is to evaluate the frequency of distant metastases and clinically relevant relapse and mortality, respectively, of aNEN (Neuroendocrine Neoplasms of the Appendix) measuring 1 - 2 cm.

The investigators hypothesize that the mortality rate of aNET (Neuroendocrine Tumors of the Appendix) measuring 1 - 2cm is less than 1%. Furthermore, the investigators hypothesize that regional lymph node metastases of aNET measuring 1 - 2 cm are clinically not relevant and are not associated with reduced survival. The investigators therefore hypothesize that oncological right-sided hemicolectomy has no impact on long-term survival after complete resection of aNET measuring 1 - 2 cm and that the malignant potential quo ad vitam of these tumors is lower than the risk of oncological hemicolectomy.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will include all patients with aNET measuring 1 - 2 cm and complete resection between 01.01.2005 and 31.12.2010 of the primary tumor.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators will include all patients with aNET measuring 1 - 2 cm and complete resection between 01.01.2005 and 31.12.2010 of the primary tumor.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Clinically relevant relapse of aNET measuring 1 - 2 cm in a population based manner | 10 years
Clinically relevant mortality of aNET measuring 1 - 2 cm in a population based manner | 10 years
Frequency of distant metastases in aNET measuring 1-2 cm | 10 years

SECONDARY OUTCOMES:
Association of histological risk factors in aNET measuring 1 - 2 cm and qualifying for oncological right-sided hemicolectomy according to ENETS guidelines with the occurrence of regional lymph node and distant metastases | 10 years
Relationship between regional lymph node metastasis and survival in patients with aNET measuring 1 - 2 cm | 10 years
Long-term survival after complete resection of aNET measuring 1 - 2 cm with or without oncological right-sided hemicolectomy | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Reto Kaderli, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- UHIBerne, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nesti C, Brautigam K, Benavent M, Bernal L, Boharoon H, Botling J, Bouroumeau A, Brcic I, Brunner M, Cadiot G, Camara M, Christ E, Clerici T, Clift AK, Clouston H, Cobianchi L, Cwikla JB, Daskalakis K, Frilling A, Garcia-Carbonero R, Grozinsky-Glasberg S, Hernando J, Hervieu V, Hofland J, Holmager P, Inzani F, Jann H, Jimenez-Fonseca P, Kacmaz E, Kaemmerer D, Kaltsas G, Klimacek B, Knigge U, Kolasinska-Cwikla A, Kolb W, Kos-Kudla B, Kunze CA, Landolfi S, La Rosa S, Lopez CL, Lorenz K, Matter M, Mazal P, Mestre-Alagarda C, Del Burgo PM, van Dijkum EJMN, Oleinikov K, Orci LA, Panzuto F, Pavel M, Perrier M, Reims HM, Rindi G, Rinke A, Rinzivillo M, Sagaert X, Satiroglu I, Selberherr A, Siebenhuner AR, Tesselaar MET, Thalhammer MJ, Thiis-Evensen E, Toumpanakis C, Vandamme T, van den Berg JG, Vanoli A, van Velthuysen MF, Verslype C, Vorburger SA, Lugli A, Ramage J, Zwahlen M, Perren A, Kaderli RM. Hemicolectomy versus appendectomy for patients with appendiceal neuroendocrine tumours 1-2 cm in size: a retrospective, Europe-wide, pooled cohort study. Lancet Oncol. 2023 Feb;24(2):187-194. doi: 10.1016/S1470-2045(22)00750-1. Epub 2023 Jan 11. PMID 36640790